CLINICAL TRIAL: NCT03288987
Title: A Phase III, Randomized, Two-armed, Triple Blinded, Parallel, Active Controlled Non-Inferiority Clinical Trial of Stivant (AryoGen Trastuzumab) Efficacy and Safety in Comparison to Avastin in Metastatic Colorectal Cancer
Brief Title: Comparing Efficacy and Safety of Stivant (AryoGen Bevacizumab) Versus Avastin in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEV.ARY.HR.94 (III)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) (Experimental): Bevacizumab+FOLFIRI-3 (irinotecan, leucovorin, and 5-FU). Bevacizumab (AryoGen) 5 mg/kg will be administered every 2 weeks.
  Interventions: Drug: Bevacizumab + FOLFIRI-3
- Bevacizumab + FOLFIRI-3 (Roche Bevacizumab) (Active Comparator): Bevacizumab+FOLFIRI-3 (irinotecan, leucovorin, and 5-FU). Bevacizumab (Avastin®) 5 mg/kg will be administered every 2 weeks.
  Interventions: Drug: Bevacizumab + FOLFIRI-3

INTERVENTIONS:
Drug: Bevacizumab + FOLFIRI-3 — Bevacizumab 5 mg/kg will be administered at day 1 every 2 weeks. Initially, it will be administered as a 90-min infusion. If the first infusion is well tolerated, the second will be delivered as a 60-min infusion, and if the 60-min infusion is well tolerated, all subsequent infusions will be given over 30 minutes. FOLFIRI-3 regimen consists of irinotecan 100 mg/m2 over 1 hour at day 1, leucovorin 400 mg/m2 at day 1 followed by a 46 hour 5-FU continuous infusion (2000 mg/m2) and irinotecan 100 mg/m2 over 1 hour on day 3 will administer. Induction treatment was administrated every 2 weeks until disease progression, unacceptable toxicities, surgical intervention, or withdrawal of consent.
  Other Names: FOLFIRI-3 = irinotecan + calcium folinate + 5-fluorouracil

SUMMARY:
This is a Phase III, randomized, two arms, double-blind (patient and assessor blinded), parallel active non inferiority controlled clinical trial with a 2:1 allocation. This trial was conducted to evaluate the efficacy and safety of bevacizumab (produced by AryoGen Pharmed) plus FOLFIRI-3 compared with bevacizumab (Avastin®) plus FOLFIRI-3 in patients with metastatic colorectal cancer (mCRC). Patients who met the following criteria could be recruited to receive the mentioned intervention randomly. Inclusion criteria: male or female aged 18-75 years, mCRC verified histologically, Having one or more bi-dimensionally measurable lesions as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria, Was not felt to be amenable to curative resection, With an (ECOG) performance status of ≤ 1, Life expectancy of longer than 3 months, Adequate organ and marrow function, May have received adjuvant therapy for primary colorectal cancer provided that at least 6 months have elapsed from the time the adjuvant therapy was concluded and recurrent disease was documented, Patients with history of hypertension must be well-controlled (blood pressure less than/equal to 150/100), on a stable regimen of anti-hypertensive therapy.

DETAILED DESCRIPTION:
This is a Phase III, randomized, two arms, double-blind (patient and assessor blinded), parallel active non inferiority controlled clinical trial with a 2:1 allocation. This trial was conducted to evaluate the efficacy and safety of bevacizumab (produced by AryoGen) plus FOLFIRI-3 compared with bevacizumab (Avastin®) plus FOLFIRI-3 in patients with metastatic colorectal cancer (mCRC). Patients who met the following criteria could be recruited to receive the mentioned intervention randomly. Inclusion criteria: male or female aged 18-75 years, mCRC verified histologically, Having one or more bi-dimensionally measurable lesions as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria, Was not felt to be amenable to curative resection, With an (ECOG) performance status of ≤ 1, Life expectancy of longer than 3 months, Adequate organ and marrow function, May have received adjuvant therapy for primary colorectal cancer provided that at least 6 months have elapsed from the time the adjuvant therapy was concluded and recurrent disease was documented, Patients with history of hypertension must be well-controlled (blood pressure less than/equal to 150/100), on a stable regimen of anti-hypertensive therapy. Exclusion criteria: Prior targeted therapy for mCRC, Radiotherapy or surgery for mCRC less than 4 weeks before random assignment, Undergone major surgical procedures or open biopsy within 28 days before the initiation of study treatment, Experienced significant traumatic injury, within 28 days before study entry, Currently using or had recently used therapeutic anticoagulants, thrombolytic therapy, chronic, daily treatment with aspirin (higher than 325 mg/daily), Proteinuria exceeding 500mg/24 h, History or presence of central nervous system metastases, Female patients who are pregnant or lactating, Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, irinotecan, 5-FU, or leucovorin, Serious non-healing wound, ulcer, or active bone fracture, Myocardial infarction within 6 months before of study enrollment, History of stroke within 6 months before of study enrollment, Unstable symptomatic arrhythmia requiring medication, Clinically significant peripheral vascular disease, Uncontrolled diabetes; Serious active or uncontrolled infection, Inability to comply with study and/or follow-up procedures. The primary endpoint is progression-free survival and overall survival, Objective Response rate, time of treatment failures, adverse events and immunogenicity will be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female aged 18-75 years at the time of signing the informed consent form.
* Have been diagnosed as mCRC verified histologically
* Having one or more bi-dimensionally measurable lesions as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria,
* Was not felt to be amenable to curative resection,
* With an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Life expectancy of longer than 3 months ( clinical assessment)
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) greater than/equal to 1,500/mm3;
  * Platelets greater than/equal to 100,000/ mm3;
  * Hemoglobin greater than/equal to 9 gm/dl (may be transfused to maintain or exceed this level);
  * Total bilirubin less than/equal to 1.5 within institutional upper limit of normal (IULN);
  * Aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) less than/equal to 2.5 times IULN, or less than/equal to 5 times IULN if known liver metastases;
* May have received adjuvant therapy for primary colorectal cancer provided that at least 6 months have elapsed from the time the adjuvant therapy was concluded and recurrent disease was documented
* Patients with history of hypertension must be well-controlled (blood pressure less than/equal to 150/100), on a stable regimen of anti-hypertensive therapy.

Exclusion Criteria:

* Prior targeted therapy for mCRC
* Radiotherapy or surgery for mCRC less than 4 weeks before random assignment.
* Undergone major surgical procedures or open biopsy within 28 days before the initiation of study treatment
* Experienced significant traumatic injury, within 28 days before study entry
* Currently using or had recently used therapeutic anticoagulants, thrombolytic therapy, chronic, daily treatment with aspirin (higher than 325 mg/daily). (Patients may have prophylactic use of low molecular weight heparin, however therapeutic use of heparin or low molecular weight heparin is not acceptable)
* Proteinuria exceeding 500mg/24 h
* History or presence of central nervous system metastases
* Female patients who are pregnant or lactating
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, irinotecan, 5-FU, or leucovorin
* Serious non-healing wound, ulcer, or active bone fracture
* Myocardial infarction within 6 months before of study enrollment;
* History of stroke within 6 months before of study enrollment;
* Clinically significant peripheral vascular disease;
* Uncontrolled diabetes; Serious active or uncontrolled infection
* Inability to comply with study and/or follow-up procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Rezvani, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (22):
- Iran (22):
  - Shafa Hospital, Ahvāz
  - Shahid Beheshti Hospital, Hamadan
  - Saba Clinic, Isfahan
  - Sheikh Mofid, Isfahan
  - Payandeh Clinic, Kermanshah
  - Shazad Clinic, Kermanshah
  - Imam Reza Hospital, Mashhad
  - Qaem Hospital, Mashhad
  - Rasool Hospital, Rasht
  - Razi Hospital, Rasht
  - Namazi Hospital, Shiraz
  - Firoozgar Hospital, Tehran
  - Imam Khomeini Hospital, Tehran
  - Imam Reza Hospital (501 Artesh), Tehran
  - Masih Daneshvari Hospital, Tehran
  - Masoud Internal Clinic, Tehran
  - Safa najafi clinic, Tehran
  - Shariati Hospital, Tehran
  - Sina Hospital, Tehran
  - Taleqani Hospital, Tehran
  - Mortazavizadeh Clinic, Yazd
  - Seyedshohada Hospital, Yazd

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezvani H, Mortazavizadeh SM, Allahyari A, Nekuee A, Najafi SN, Vahidfar M, Ghadyani M, Khosravi A, Qarib S, Sadeghi A, Esfandbod M, Rajaeinejad M, Rezvani A, Hajiqolami A, Payandeh M, Shazad B, Anjidani N, Meskinimood S, Alikhasi A, Karbalaeian M, Salari S. Efficacy and Safety of Proposed Bevacizumab Biosimilar BE1040V in Patients With Metastatic Colorectal Cancer: A Phase III, Randomized, Double-blind, Noninferiority Clinical Trial. Clin Ther. 2020 May;42(5):848-859. doi: 10.1016/j.clinthera.2020.03.009. Epub 2020 Apr 22. PMID 32334845
- See also: Efficacy and Safety of Proposed Bevacizumab Biosimilar BE1040V in Patients With Metastatic Colorectal Cancer: A Phase III, Randomized, Double-blind, Noninferiority Clinical Trial — http://pubmed.ncbi.nlm.nih.gov/32334845/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Started | 82 | 44
Patients Receiving Medication | 80 | 44
Completed | 72 (Per protocol population) | 40 (Per protocol population)
Not Completed | 10 | 4
Not completed — Protocol Violation | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab) | Total
Number analyzed (Participants) | 82 | 44 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.26 (11.94) | 56.27 (13.12) | 56.26 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 15 | 46
  Male | 51 | 29 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 82 | 44 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the first date of documentation progression (per investigator assessment) or death as a result of any cause.
Time Frame: PFS was measured from the start of chemotherapy to the date of disease progression or to the date of death if no progression whichever came first, assessed up to 12 months
Population: The population assessable for PFS was per protocol.
Measure: Median (Standard Error); unit: Day
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Number analyzed (Participants) | 72 | 40
Day | 232 (NA) — The median has been obtained from the KM (SPSS) using the 50th percentile and the standard error from the 45th percentile. However, it was not possible to compute the standard error (45th percentile) for AryoGen Bevacizumab because the data from the survival function did not reach the 45th percentile. This was possible for the Bevacizumab of Roche. Data should be seen in the publication of study results. | 210 (12.21)
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) vs Bevacizumab + FOLFIRI-3 (Roche Bevacizumab); Test type: Non-Inferiority — Noninferiority was declared by comparing the 90% CI for the hazard ratio (HR) of the AryoGen Pharmed Bevacizumab to the reference product (Roche Bevacizumab) to the point-estimate margin and was based on the synthesis method; p = 0.47, Regression, Cox; Upper limit of CI is lower than the noninferiority margin (1.44); Hazard Ratio (HR) = 0.79, 90% CI 2-sided [0.46 to 1.35] — The 90 % CI based on synthesis method is (0.45,1.38). In HR calculation, the AryoGen Pharmed Bevacizumab to Roche Bevacizumab was reported. (reference group was Roche Bevacizumab)

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival OS was defined as the time from date of randomization to date of death due to any cause
Time Frame: Up to 12 months
Population: ITT population was used in this outcome analysis. The probability of overall survival in this study was higher than 50% in one year, so the calculation of median was not applicant.
  The number of death in both arms is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Number analyzed (Participants) | 82 | 44
Participants | 30 | 17
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) vs Bevacizumab + FOLFIRI-3 (Roche Bevacizumab); Test type: Other; p = 0.99, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.55 to 1.80] — In HR calculation, the AryoGen Pharmed Bevacizumab to Roche Bevacizumab was reported. (reference group was Roche Bevacizumab)

3. Secondary Outcome: Objective Response Rate
Description: Tumor response was defined as partial and complete responses, according to the RECIST criteria ( version 1.1). The definitions were as follows: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), decrease of at least 30% in the lesion that has the largest diameter; Objective Response Rate (ORR) = CR + PR.
Time Frame: Up to 12 months
Population: Both baseline imaging and imaging at the time of withdrawal, could not be gathered in all patients. So ORR could be reported in the mentioned population in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Number analyzed (Participants) | 42 | 23
Participants | 17 | 5
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) vs Bevacizumab + FOLFIRI-3 (Roche Bevacizumab); Test type: Other; p = 0.17, Fisher's Exact Test

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from the date of randomization to the date of each of the following,
  * The treatment modalities did not destroy or modify the cancer cells,
  * The tumor either became larger (disease progression) or stayed the same size after treatment,
  * Death due to any cause,
  * Discontinuation of treatment
Time Frame: Up to 12 months
Measure: Median (Standard Error); unit: Day
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Number analyzed (Participants) | 80 | 44
Day | 73 (9.39) | 73 (9.12)
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) vs Bevacizumab + FOLFIRI-3 (Roche Bevacizumab); Test type: Other; p = 0.59, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.76 to 1.61] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Incidence of the Adverse Events
Description: Safety was assessed on the basis of reports of adverse events, laboratory-test results, and vital sign measurements. Adverse events were categorized According to the Common Toxicity Criteria of the National Cancer Institute, version 5.0, in which a grade of 1 indicates mild adverse events, a grade of 2 moderate adverse events, a grade of 3 serious adverse events, and a grade of 4 life-threatening adverse events
Time Frame: Up to 12 months
Population: A total of 124 patients were analyzed for AEs. since two patients did not receive study medication and were not included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Number analyzed (Participants) | 80 | 44
Participants | 76 | 44
Statistical Analysis 1: Comparison: Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) vs Bevacizumab + FOLFIRI-3 (Roche Bevacizumab); Test type: Other; p > 0.05, Fisher's Exact Test

6. Secondary Outcome: Number of Positive Anti-drug Antibody (ADA) Samples Among Patients (Immunogenicity)
Description: Anti-drug antibody assessment
Time Frame: Up to 12 months
Population: Positive ADA was reported in two patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
Number analyzed (Participants) | 82 | 44
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The Safety Population included patients who received at least one dose of the investigational medicines. The different definition of the ITT (all patients who were randomized) should explain the inconsistency across the All-cause Mortality ( ITT population: 82 patients in the group treated with Bevacizumab AryoGen and 44 patients in the group Bevacizumab Roche) and SAE/ Other AE (Safety Population: 80 patients in the group Bevacizumab AryoGen and 44 patients in the group Bevacizumab Roche).
Arm/Group | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 30/82 | 17/44
Serious Adverse Events (participants affected / at risk) | 31/80 | 17/44
Other Adverse Events (participants affected / at risk) | 75/80 | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) (N=80) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab) (N=44)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 25 (25) | 15 (15)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Opioid abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Perforation (General disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + FOLFIRI-3 (AryoGen Pharmed Bevacizumab) (N=80) | Bevacizumab + FOLFIRI-3 (Roche Bevacizumab) (N=44)
Anaemia (Blood and lymphatic system disorders) | 62 (131) | 37 (76)
Leukopenia (Blood and lymphatic system disorders) | 22 (42) | 19 (25)
Neutropenia (Blood and lymphatic system disorders) | 25 (46) | 15 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (3) | 1 (2)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diabetic foot (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 43 (67) | 28 (50)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (10) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (27) | 6 (7)
Proctalgia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Febrile neutropenia (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (3) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 22 (33) | 9 (13)
Aspartate aminotransferase increased (Investigations) | 24 (34) | 9 (14)
Blood bilirubin increased (Investigations) | 10 (16) | 9 (9)
Blood creatinine increased (Investigations) | 5 (10) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 20 (36) | 11 (15)
Lymphocyte count abnormal (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (13) | 3 (5)
Platelet count decreased (Investigations) | 10 (10) | 7 (7)
Weight decreased (Investigations) | 9 (10) | 6 (6)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6) | 6 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysphonia (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Tachyphrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 13 (25) | 7 (8)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 18 (32) | 12 (15)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteritis (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhoids (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 11 (19) | 5 (8)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03288987/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03288987/Prot_ICF_001.pdf